CLINICAL TRIAL: NCT05190133
Title: An Open-label, Multiple-dosing, Two-arms, One-sequence Study to Evaluate the Safety and Pharmacokinetics After Co-administration of UIC201601 and UIC201602 in Healthy Male Volunteers
Brief Title: Drug-drug Interaction Study Between UIC201601 and UIC201602
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: KUP-UI018-101
Record Dates: First submitted 2021-12-22; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental)
  Interventions: Drug: UIC201602 and co-administration of UIC201601 and UIC201602
- Treatment B (Experimental)
  Interventions: Drug: UIC201601 and co-administration of UIC201601 and UIC201602

INTERVENTIONS:
Drug: UIC201602 and co-administration of UIC201601 and UIC201602 — * UIC201602 4 Cap/day for 14 days
  * Wash out 21 days
  * UIC201601 4 Tab + UIC201602 4 Cap / day for 14 days
  Arms: Treatment A
Drug: UIC201601 and co-administration of UIC201601 and UIC201602 — * UIC201601 4 Tab/day for 7 days
  * Wash out 14 days
  * UIC201601 4 Tab + UIC201602 4 Cap / day for 14 days
  Arms: Treatment B

SUMMARY:
An open-label, multiple-dosing, two-arms, one-sequence study to evaluate the safety and pharmacokinetics after co-administration of UIC201601 and UIC201602 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose body weight over 55 kg and ranged ± 20% of calculated Ideal Body Weight;
* Subjects without congenital disease, chronic disease, symptom or any clinical significance of a physical examination and questionnaires;
* Subjects judged as healthy by laboratory tests including blood haematology, biochemistry, urinalysis and serologic tests;
* Subjects able to read and understand a written informed consent, and willing to participate in the study.

Exclusion Criteria:

* Subjects with clinically significant symptoms or medical histories on liver, kidney, neuronal system, respiratory system, haematology, oncology, mental illness and particularly cardiovascular system (hypertension, angina, heart failure, myocardial infarction, etc.) or endocrine system (diabetes, hyperlipidemia, etc);
* Subjects with chronic disease which might affect drug absorption, distribution, metabolism and elimination;
* Subjects with a medical history of clinically significant hypersensitivity or hypersensitivity to the drug-containing atorvastatin or HMG-CoA reductase inhibitor;
* Subjects with a medical history of clinically significant hypersensitivity or hypersensitivity to omega-3 or fish;
* Subject with generic metabolic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption;
* etc.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-28 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics(AUCss,τ) of UIC201602 | 0 hour to 24 hours after Day 14 and Day 49 administration
  Area under the serum drug concentration-time curve within a dosing interval at steady state
Plasma pharmacokinetics(Css,max) of UIC201602 | 0 hour to 24 hours after Day 14 and Day 49 administration
  Maximum concentration of drug in serum at steady state
Plasma pharmacokinetics(AUCss,τ) of UIC201601 | 0 hour to 24 hours after Day 7 and Day 35
  Area under the serum drug concentration-time curve within a dosing interval at steady state
Plasma pharmacokinetics(Css,max) of UIC201601 | 0 hour to 24 hours after Day 7 and Day 35
  Maximum concentration of drug in serum at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Janghee Hong, M.D.,Ph.D., Principal Investigator — Chungnam National University Hospital

IPD SHARING:
Plan to Share IPD: No